CLINICAL TRIAL: NCT01221051
Title: A Comparison of Active and Expectant Management of the Third Stage of Labor
Brief Title: Third Stage of Labor a Swedish Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VGFOUGSB-8290
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Childbirth
Keywords: third stage of labor,oxytocics, postpartum hemorrhage,
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxytocin (Active Comparator): early cord clamping, administration of oxytocin 10 IU i.v, controlled cord traction, uterine massage after placenta expulsion
  Interventions: Procedure: active management of the third stage of labor
- saline solution (Placebo Comparator): early cord clamping, wait for signs of placenta detachment, encourage the woman to push out placenta by her own effort, uterine massage after placenta expulsion
  Interventions: Procedure: expectant management of the third stage of labor

INTERVENTIONS:
Procedure: active management of the third stage of labor — early cord clamping, administration of oxytocin 10 IU, controlled cord traction, uterine massage after placenta expulsion
  Other Names: AMTSL
  Arms: oxytocin
Procedure: expectant management of the third stage of labor — early cord clamping, administer saline solution 2 mL i.v,wait for signs of placenta detachment, encourage the woman to push ot placenta by her own effort, uterine massage after placenta expulsion
  Other Names: EMTSL
  Arms: saline solution

SUMMARY:
The purpose with this study was to compare blood loss and women's experience of afterpains during the third stage when handled with active or expectant management of the third stage of labour.

Hypothesis 1. To detect a 5% difference (15% vs 10%) in blood loss >1000 mL between the two groups with 80% power (α=0.05), at least 726 subjects were required in each group.

Hypothesis 2. Afterpains are more pronounced in active compared to expectant management during the third stage of labour

DETAILED DESCRIPTION:
Management of the third stage of labour has been focus for investigation during decades and active management of the third stage of labour (AMTSL)has been recommended in all women giving birth vaginally at hospitals. In Sweden the recommendation has been to give an injection of oxytocin immediately after birth of the neonate but not the entire AMTSL procedure.

Women in labour were asked to participate voluntarily when entering the hospital and after acceptance they were randomised to either active or expectant management of the third stage of labour(EMTSL).

AMTSL included:

* Early cord clamping
* 10 UI oxytocin i.v
* controlled cord traction
* uterine massage after placenta expulsion

EMTSL included:

* early cord clamping
* 2 mL saline solution i.v
* wait for signs of placenta detachment
* encourage the women to push out placenta by her own effort
* uterine massage after placenta expulsion

All blood was measured by weighing bed pads and sanitary towels up to two hours postpartum Assessment of afterpains was performed by a Visual Analogue Scale (VAS) and the Pain-o-meter (POM-WDS) two hours after the delivery of placenta, and the day after childbirth.

ELIGIBILITY:
Inclusion Criteria:

* healthy women with normal pregnancies
* gestational age of 34+0 - 43+0 weeks
* singleton, cephalic presentation
* expected vaginal birth

Exclusion Criteria:

* non Swedish-speaking
* previous PPH >1000 mL
* elective Caesarean section
* pre-eclampsia
* grand multiparity (≥5)
* intrauterine fetal death

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
blood loss | blood loss measured up to two hours post partum
  All blood was collected and measured from delivery of the infant and two hours after.

SECONDARY OUTCOMES:
afterpains | at two hours postpartum and the day after delivery
  Women assessed their afterpains at two hours and the day after delivery

CONTACTS AND LOCATIONS:
Overall Officials: elisabeth jangsten, Principal Investigator — Sahlgrenska academy, University of Gothenburg